CLINICAL TRIAL: NCT05307796
Title: Incorporating Strategy Training Into Naming Treatment to Improve Generalization in Aphasia
Brief Title: Incorporating Strategy Training Into Naming Treatment in Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MGH Institute of Health Professions (Other)
Collaborators: LSVT Global (Unknown)
Responsible Party: Principal Investigator, Sofia Vallila Rohter, Associate Professor, MGH Institute of Health Professions
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021P000705
Record Dates: First submitted 2022-03-22; First posted 2022-04-01 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Aphasia
Keywords: Aphasia; Naming; Circumlocution
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Semantic Feature Analysis plus metacognitive strategy training (Experimental): Participants attend three treatment sessions per week for eight weeks. Treatment sessions include: strategy education (participants learn about anomia, circumlocution, and circumlocution's purpose), Semantic Feature Analysis plus strategy application (participants build self-awareness and practice circumlocution), and strategy debriefing (participants reflect and receive feedback on their performance, and generate scenarios in which they could use the strategy in everyday life).
  Interventions: Behavioral: Strategy training

INTERVENTIONS:
Behavioral: Strategy training — The strategy training of focus in this study is metacognitive strategy training intended to build awareness of naming and methods to overcome instances of difficult naming. Strategy training involves (a) teaching the participant to identify instances in which they are unable to name objects, (b) learn a 6-feature framework (e.g. group, use, action) that has been identified to support semantic feature activation in aphasia, (c) learn and practice strategies to utilize the framework in instances of word finding difficulty

SUMMARY:
This study incorporates metacognitive strategy training into semantic feature analysis treatment. Semantic feature analysis treatment has a strong evidence base and capacity to improve word retrieval by encouraging circumlocution. Circumlocution facilitates self-cued naming and assists listener comprehension when naming fails. However, semantic feature analysis treatment does not include direct techniques to teach patients with aphasia to generalize the use of semantic feature analysis treatment's circumlocution procedure. Therefore, this study proposes that combining semantic feature analysis treatment and metacognitive strategy training will stimulate the semantic system and increase patients with aphasias' use of circumlocution across divergent contexts.

This study aims to measure the treatment's effect on naming accuracy for trained and untrained items. The study also aim to measure the treatment's effect on people with aphasias' knowledge of the strategy components and changes in verbalizations during retrieval attempts. The central hypothesis is that strategy training will increase patients with aphasias' explicit knowledge about circumlocution and enable them to use it to (1) self-facilitate naming, and (2) produce more informative connected speech.

DETAILED DESCRIPTION:
Every 40 seconds, someone in the United States suffers from a stroke. Approximately 25% of stroke survivors acquire aphasia, a communication disorder that can result in a partial or total loss of spoken and written language ability, which significantly and negatively impacts quality of life and societal participation. The ability to verbally label objects, referred to as 'naming' in the literature, is impaired in all patients with aphasia. Naming is, therefore, a common focus of treatment. Naming treatments improve people with aphasias' naming ability for items that are directly trained during therapy. However, these same treatments face two critical limitations: (1) inconsistent generalization to untrained items, and (2) little to no generalization to spontaneous, connected speech. As it is impossible to train the entire universe of objects during a patient's course of therapy, generalization of gains beyond what is trained in therapy is crucial.

Recent work shows that patients with aphasias' learning success depends on their ability to develop optimal strategies that support learning, but that they do not develop these strategies independently. There is also evidence that through explicit strategy training, patients with aphasia can learn to implement and generalize the use of strategies that are known to support learning, and carry over their use across multiple environments. As such, it is predicted that naming treatment outcomes would be greatly improved by incorporating strategy training into treatment.

This study proposes to incorporate strategy training into naming treatment to improve generalization. Circumlocution, a verbal behavior in which patients with aphasia describe an object's features if they are unable to name it, is known to facilitate naming and assist listener comprehension. Semantic Feature Analysis is a well-regarded naming treatment thought to encourage circumlocution. Semantic Feature Analysis treatment does not include direct techniques that teach patients with aphasia how to generalize the use of the treatment's circumlocution procedure. In fact, no studies have explicitly trained patients with aphasia how to use the circumlocution procedure they learn in Semantic Feature Analysis treatment during everyday communication. Rather, it is assumed that patients with aphasia will implicitly learn how to use the procedure, through repeated practice and habituation alone. This study proposes that strategy training is the integral missing piece that will successfully result in people with aphasias' generalized application of the semantic feature analysis procedure.

The objective of the proposed research is to determine whether naming treatment that incorporates strategy training results in people with aphasias' increased use of circumlocution. The central hypothesis is that strategy training will increase patients with aphasias' explicit knowledge about circumlocution and enable them to use it to (1) self-facilitate naming, and (2) produce more informative connected speech. It is predicted that increased use of circumlocution will result in generalization at both the impairment level (naming) and participation level (effective communication).

ELIGIBILITY:
Inclusion criteria:

* Experienced a single left-hemisphere stroke,
* Have aphasia due to stroke,
* Be in the chronic stages of their aphasia, at least 6 months post onset of stroke.
* Be between the ages of 18 and 89 years of age, and
* Be a proficient English speaker,
* Have no history of neurodegenerative disease, motor speech disorder, significant mental illness, psychiatric disorder, drug/alcohol abuse, or neurological condition that could influence their cognitive, language, and memory systems.

Exclusion criteria:

* Experienced multiple strokes;
* Be in the acute stage of their aphasia, <6 months post onset of stroke;
* Have a diagnosis of neurodegenerative disease, significant mental illness, psychiatric disorder, drug/alcohol abuse, or neurological condition that could influence cognitive, language, and memory systems

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
Naming accuracy | Change from baseline at 6 months
  Number of pictures named accurately when looking at a series of 176 object pictures
Strategy Use | Change from baseline at 6 months
  Number of instances of circumlocution in moments of naming difficulty when looking at a series of 176 object pictures
Strategy Knowledge | Change from baseline at 6 months
  Number of strategy components (out of 6) participants identify (verbally or gesturally) independently

SECONDARY OUTCOMES:
Content Information Units | Change from baseline at 6 months
  Number of content information units (CIUs) in connected speech samples when describing pictures and telling stories.

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Vallila Rohter, PhD, Principal Investigator — MGH Institute of Health Professions
Locations (1):
- MGH-Institute of Health Professions, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators will share de-identified data sets, statistical analysis codes and experimental set-ups with interested researchers, educators or clinicians. Materials generated under the project will be disseminated in accordance with NIH policies.
Time Frame: Data requests can be submitted starting 9 months after article publication and will be made accessible for up to 24 months
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-03): https://cdn.clinicaltrials.gov/large-docs/96/NCT05307796/Prot_SAP_000.pdf